CLINICAL TRIAL: NCT05513625
Title: A Single-center, Open-label, 2-period Fixed-sequence Phase I Trial to Evaluate the Effect of Esomeprazole on the Pharmacokinetics of Pritelivir
Brief Title: Potential Influence of Esomeprazole on the Pharmacokinetics of Pritelivir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AiCuris Anti-infective Cures AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: AIC316-03-I-01
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Results first posted 2023-09-15 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2022-09

CONDITIONS: HSV Infection
MeSH Terms: conditions — Herpes Simplex | interventions — pritelivir

STUDY DESIGN:
Intervention Model Description: Sequence for all subjects:
  Treatment 1: single dose of 100 mg PTV followed by Wash out period (4weeks) followed by Treatment 2: single dose of 100 mg PTV Day 1 and 40 mg/day ESO from Day -3 to Day 1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 100 mg pritelivir (Experimental): Single dose 100 mg pritelivir (PTV) administered day 1
  Interventions: Drug: Pritelivir
- 40 mg qd ESO and 100 mg pritelivir (Experimental): 40 mg qd ESO Day -3 to Day1. Single dose of 100 mg PTV on Day 1
  Interventions: Drug: ESO and pritelivir

INTERVENTIONS:
Drug: Pritelivir — oral administration
  Arms: 100 mg pritelivir
Drug: ESO and pritelivir — oral administration
  Arms: 40 mg qd ESO and 100 mg pritelivir

SUMMARY:
To investigate the effect of esomeprazole (ESO) on the pharmacokinetics of pritelivir (PTV), and to investigate the safety and tolerability of PTV.

DETAILED DESCRIPTION:
This was a single-center, open-label, 2-period, fixed-sequence Phase 1 trial in 16 healthy adult male and female subjects (at least 7 subjects per sex). In the first period, subjects received treatment 1 (T1; single dose of 100 mg PTV on Day 1). In the second period, subjects received treatment 2 (T2: 40 mg qd ESO from Day -3 to Day 1 followed by a single dose of 100 mg PTV on Day 1). The wash-out period between PTV administrations in T1 and T2 was at least 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects had to have the ability to understand and sign written informed consent, which had to be obtained prior to any trial-related procedures being completed;
2. Healthy male and female subjects of any ethnic origin, aged between 18 and 45 years (inclusive) assessed as healthy based on a pre-trial examination including medical history, physical examination, blood pressure, pulse rate, electrocardiogram (ECG) assessment, and clinical laboratory results.
3. Female subjects of non-childbearing potential had to be either surgically sterile (hysterectomy, bilateral tubal ligation, salpingectomy, and/or bilateral oophorectomy at least 26 weeks prior to Screening) or postmenopausal, defined as spontaneous amenorrhea for at least 2 years, with follicle-stimulating hormone (FSH) in the postmenopausal range at Screening based on the central laboratory's ranges.
4. Female subjects of childbearing potential (ie, ovulating, premenopausal, and not surgically sterile) and all male subjects had to use a medically accepted contraceptive regimen during their participation in the trial and for 90 days after the last administration of trial drug. Medically accepted contraceptive methods were defined as those with 90% or greater efficacy.

   Acceptable methods of contraception for male subjects enrolled in the trial included the following:
   * Condoms with spermicide.
   * Surgical sterilization of the subject at least 26 weeks prior to Screening (vasectomy).

   Acceptable methods of contraception for female subjects enrolled in the trial included the following, (the subject had to choose two of the following [a single barrier method alone or abstinence alone was not acceptable]):
   * Condoms with spermicide.
   * Intrauterine device for at least 12 weeks prior to Screening.
   * Hormonal contraception (oral, implant, injection, ring, or patch) for at least 12 weeks prior to Screening.
   * Diaphragm used in combination with spermicide.
5. Male subjects had to agree to abstain from sperm donation and not plan to father a child (including sperm donation) through 90 days after administration of the last dose of trial drug.
6. In women: a negative serum beta-human chorionic gonadotropin (β-HCG) test at Screening and negative urine β-HCG test at Admission in each Treatment Period.
7. Subject agreed to pharmacogenetic blood sampling.
8. Normal body weight as evidenced by a Body Mass Index (BMI) ≥18.0 and ≤32.0 kg/m2, and a body weight ≥50.0 kg at Screening.
9. Subjects had to have a negative test result for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCVAb), and human immunodeficiency virus (HIV) at Screening;
10. Subjects had to have negative urine tests for drugs of abuse (metamphetamines, amphetamines, 3,4-Methylendioxyamphetamin (MDMA), barbiturates, benzodiazepines, cannabinoids, opioids, cocaine and tricyclic antidepressants) and negative breath alcohol tests at Screening and Admission in each Treatment Period.

Exclusion criteria:

1. History or current evidence of clinically relevant allergies or idiosyncrasy to drugs or food
2. History of allergic reactions to any active or inactive ingredient(s) of the trial medication(s)
3. History or current evidence of any clinically relevant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, hematological, endocrinological, metabolic, neurological, psychiatric, or other disease suspected to influence pharmacokinetics or safety of PTV
4. History of malignancy
5. Resting pulse rate after 5 minutes in supine position at Screening and Day -1 of Treatment Period 1: <45 or >100 beats per minute (bpm), if out of range, up to one repeat assessment was allowed
6. Resting blood pressure after 5 minutes in supine position at Screening and Day -1 of Treatment Period 1: systolic blood pressure <90 or >145 mmHg diastolic blood pressure <40 or >95 mmHg, if out of range, up to one repeat assessment was allowed
7. ECG abnormalities of clinical relevance (eg, QTc according to Fridericia: QTc >450 ms in males and >470 ms in females; PR ≥220 ms)
8. Febrile or infectious illness within 5 days prior to administration of Investigational Medicinal Product
9. Clinically relevant abnormalities in clinical chemical, hematological or any other laboratory variables
10. Chronic or clinically relevant acute infections
11. Diagnosed to be COVID-19 positive by polymerase chain reaction (PCR) testing (SARS-CoV-2 RT-PCR positive) of a respiratory specimen (preferably a nasopharyngeal swab) on Day -2 of Treatment Period 1
12. Subject was lactating or breastfeeding
13. Use of any medication (incl. over-the-counter [OTC] medication) within 2 weeks before first drug administration or within less than 10 times the elimination half-life of the respective drug, or anticipated concomitant medication during the treatment periods. Use of hormonal contraceptives was allowed. Single intake of a drug may have been accepted if judged by the Investigators to have no clinical relevance and no relevance for the trial objectives. Limited amounts of acetaminophen were allowed to treat painful intercurrent adverse events (eg, headache, migraine).
14. Consumption of any (eg, CYP1A2, CYP3A4) enzyme inducing or inhibiting aliments and beverages (eg, but not limited to broccoli, Brussels sprout, grapefruit, grapefruit juice, Seville orange, star fruit, tonic water, bitter lemon etc.) within 2 weeks prior to the Screening (Pre-trial examination)
15. Consumption of methylxanthine-containing beverages or food (coffee, tea, cola, chocolate, "powerdrinks") from 24 hours before PTV dosing on Day 1 until release from the clinic on Day 5 of each period
16. Consumption of alcohol and tobacco products within 48 hours prior to admission to the clinic until discharge of each period
17. Vegetarian diet or other dietary habits which would have precluded the subject's acceptance of standardized meals
18. Diseases or surgery of the gastrointestinal tract which may have interfered with drug absorption (note: this was not applicable for minor abdominal surgery such as eg, appendectomy and herniotomy)
19. Receipt of any Investigational Medicinal Product (IMP) within a time period equal to 10 half-lives of the product, if known, or a minimum of 30 days prior to trial drug administration.
20. Blood donation or loss of 550 mL or more within the last 30 days before start of Screening (Pre-trial examination)
21. Smoking of more than 10 cigarettes/cigars/pipes per Day and/or inability to refrain from smoking during confinement
22. Intake of more than 12 units of alcohol per week (one unit of alcohol equals approximately 250 mL of beer, 100 mL of wine or 35 mL of spirits)
23. Had any finding that, in the view of the Investigator, would have compromised the subject's safety requirements

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2020-10-13 (Actual); Study Completion 2020-10-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medpace Clinical Pharmacology, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 16 subjects enrolled in PTV 100 mg (T1), 15 completed. The 15 completed were enrolled into ESO 40 mg/PTV 100 mg (T2)
Groups:
- 100 mg Pritelivir / 40 mg qd ESO and 100 mg Pritelivir: Single dose 100 mg pritelivir (PTV) administered day 1
  Pritelivir: oral administration
  40 mg qd ESO Day -3 to Day1. Single dose of 100 mg PTV on Day 1
  ESO and pritelivir: oral administration
Period: Overall Study
Arm/Group | 100 mg Pritelivir / 40 mg qd ESO and 100 mg Pritelivir
Started | 16
Completed | 15
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Safety Set
Arm/Group | 100 mg Pritelivir / 40 mg qd ESO and 100 mg Pritelivir
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.6 (8.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: PK - Cmax
Description: Cmax - the maximum observed plasma concentration
Time Frame: 15 days
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- 100 mg Pritelivir: Single dose 100 mg pritelivir (PTV) administered on Day 1
  Pritelivir: oral administration
Arm/Group | 100 mg Pritelivir | 40 mg qd ESO and 100 mg Pritelivir
Number analyzed (Participants) | 16 | 15
ng/mL | 1102 (421) | 282 (141)

2. Primary Outcome: PK - AUC(0-infinity) and AUC(0-last)
Description: AUC0-∞ - area under the analyte vs time concentration curve from time of administration up to infinity, calculated as AUC0-∞ = AUC0-last + (Clast / λz)
  AUC0-last - area under the analyte vs. time concentration curve from time of administration up to the time of the last quantifiable concentration, calculated by linear up/ln down summation
Time Frame: 15 days
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | 100 mg Pritelivir | 40 mg qd ESO and 100 mg Pritelivir
Number analyzed (Participants) | 15 | 15
ng*h/mL
  AUC(0-last) | 67599 (22012) | 28325 (11071)
  PK - AUC(0-infinity) | 69140 (22147) | 29404 (11447)

3. Secondary Outcome: PK - Tmax and Tlag
Description: tmax - time to reach the maximal observed analyte concentration and tlag - time period between the time of dosing and the time of the first measurable concentration
Time Frame: 15 days
Measure: Median (Full Range); unit: hours
Arm/Group | 100 mg Pritelivir | 40 mg qd ESO and 100 mg Pritelivir
Number analyzed (Participants) | 16 | 15
hours
  tmax | 3.00 [0.50 to 10.00] | 8.00 [0.75 to 48.00]
  tlag | 0.00 [0.00 to 0.25] | 0.00 [0.00 to 0.25]

4. Secondary Outcome: PK - λz
Description: λz - the apparent terminal elimination rate constant, determined by linear regression of terminal points of the ln-linear analyte concentration-time curve
Time Frame: 15 days
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | 100 mg Pritelivir | 40 mg qd ESO and 100 mg Pritelivir
Number analyzed (Participants) | 15 | 15
1/h | 0.0106 (0.0020) | 0.00970 (0.0018)

5. Secondary Outcome: PK t1/2z
Description: t1/2z - the apparent terminal elimination half-life calculated as: t1/2z = 0.693 / λz
Time Frame: 15 days
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 100 mg Pritelivir | 40 mg qd ESO and 100 mg Pritelivir
Number analyzed (Participants) | 15 | 15
hours | 67.7 (12) | 73.7 (13)

6. Secondary Outcome: PK - CL/F
Description: CL/F - total apparent clearance of drug following single dose e.v. administration calculated as: CL/F = Dose / AUC0-∞
Time Frame: 15 days
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | 100 mg Pritelivir | 40 mg qd ESO and 100 mg Pritelivir
Number analyzed (Participants) | 15 | 15
L/h | 1.58 (0.46) | 3.93 (1.6)

7. Secondary Outcome: V d/F
Description: V d/F - apparent volume of distribution after a single dose e.v. administration calculated as Vd/F = Dose e.v. / (λz * AUC0-∞)
Time Frame: 15 days
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 100 mg Pritelivir | 40 mg qd ESO and 100 mg Pritelivir
Number analyzed (Participants) | 15 | 15
L | 157 (63) | 432 (231)

ADVERSE EVENTS:
Time Frame: 32 days
Arm/Group | 100 mg Pritelivir | 40 mg qd ESO and 100 mg Pritelivir
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 2/16 | 4/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 100 mg Pritelivir (N=16) | 40 mg qd ESO and 100 mg Pritelivir (N=15)
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Tooth impacted (Gastrointestinal disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-16): https://cdn.clinicaltrials.gov/large-docs/25/NCT05513625/Prot_SAP_000.pdf